CLINICAL TRIAL: NCT06510738
Title: Prediction of Non-sentinel Lymph Node Metastatic Status of Breast Cancer Based on Pathology-MRI Images and Artificial Intelligence
Brief Title: Prediction of Non-sentinel Lymph Node Metastatic Status of Breast Cancer Based on Pathology-MRI Images
Status: Not yet recruiting | Type: Observational
Sponsor: Yunnan Cancer Hospital (Other)
Collaborators: Affiliated Cancer Hospital of Shantou University Medical College (Other)
Responsible Party: Sponsor
Other Study IDs: KYLX2024-128
Record Dates: First submitted 2024-07-14; First posted 2024-07-19 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer; Artificial Intelligence; Lymph Node Metastasis; Digital Pathology
MeSH Terms: conditions — Breast Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to develop an artificial intelligence model based on pathology and magnetic resonance imaging (MRI) images to predict the metastatic status of non-sentinel lymph nodes in patients with breast cancer sentinel lymph node metastasis. The main questions it aims to answer are:

Can an artificial intelligence model based on MRI images of breast cancer patients predict the non-sentinel lymph node metastatic status in patients with breast cancer sentinel lymph node metastasis?

Can an artificial intelligence model based on intraoperative frozen section images of sentinel lymph nodes in breast cancer patients predict the non-sentinel lymph node metastasis status in patients with sentinel lymph node metastasis from breast cancer?

Can artificial intelligence models based on preoperative MRI and intraoperative frozen section images of sentinel lymph nodes in breast cancer patients predict the non-sentinel lymph node metastatic status in patients with sentinel lymph node metastasis from breast cancer?

Researchers will retrospectively and prospectively collect preoperative MRI and intraoperative sentinel lymph node section images from breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary breast cancer
2. Positive sentinel lymph node biopsy and axillary lymph node dissection.
3. No neoadjuvant chemotherapy, radiotherapy or ablation prior to surgery.
4. MRI within 3 weeks prior to surgery.

Exclusion Criteria:

1. recurrent breast cancer or history of surgery or radiation therapy in the axilla
2. Inflammatory breast cancer
3. Bilateral breast cancer or metastatic breast cancer
4. previous or current history of other malignant tumors
5. Sentinel lymph node count > 5

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators plan to retrospective collect 700 patients with breast cancer and prospective collect 150 patients with breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Non-sentinel lymph node metastatic status | 2024-2025
  metastasis or non-metastasis
Accuracy, Sensitivity, Specificity，Area under the curve | 2024-2025
  The performance of predicting non-sentinel lymph node metastatic status
Positive predictive value，Negative predictive value | 2024-2025
  The performance of predicting non-sentinel lymph node metastatic status